CLINICAL TRIAL: NCT04412837
Title: The Use of Cannabinoid Patch for Knee Osteoarthritis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Inadequate funding
Sponsor: Northwell Health (Other)
Collaborators: Solace Brands, Inc. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-0048
Record Dates: First submitted 2020-05-21; First posted 2020-06-02 (Actual); Last update posted 2023-01-19 (Actual); Status verified 2023-01

CONDITIONS: Knee Osteoarthritis; CBD; Osteoarthritis
Keywords: Cannabidiol
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: This will be a randomized double blinded parallel group clinical trial to determine safety and efficacy of 35mg CBD patch vs placebo patch in patients with knee osteoarthritis.
Who Masked: Participant, Care Provider, Investigator
Masking Description: Patients, treating physician, and assessors will be blinded to study group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBD Patch (Experimental): Topical CBD patch to be worn for 24 hours and changed daily for the course of 4 weeks.
  Interventions: Drug: Topical CBD Patch
- Control Patch (Placebo Comparator): Control placebo patch to be worn for 24 hours and changed daily for the course of 4 weeks.
  Interventions: Other: Placebo Patch

INTERVENTIONS:
Drug: Topical CBD Patch — 35 mg CBD patch
  Arms: CBD Patch
Other: Placebo Patch — Identical patch without active ingredient.
  Arms: Control Patch

SUMMARY:
This randomized, double-blind 2-arm parallel group study to determine the efficacy of a cannabinoid (CBD) patch on reducing pain in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
The aim of this study is to determine the efficacy of cannabinoid (CBD) patch on reducing pain and improving functional status in patients with knee osteoarthritis (OA). The investigators hypothesize that the use of CBD patch will provide superior pain relief to placebo patch. This will be a randomized, double-blind 2-arm parallel group study in 74 male and female subjects with pain from knee osteoarthritis. Site staff will document the patient's prior treatment for knee osteoarthritis and once the diagnosis has been made, they will be offered to enroll in the study.

After randomization, patients will either be prescribed CBD patch to be used topically for diagnosed knee osteoarthritis versus placebo patch. It will be performed at one site, the physician's office. The study coordinator will be in charge of keeping track of the different patches and all other study personnel and patients will be blinded to the treatment arm. The statistician will conduct the randomization. He will be unblinded and assign participant numbers.

Patients will be diagnosed in an office setting for knee osteoarthritis based on radiographs using the Kellgren Lawrence classification. It is the standard of care to obtain orthogonal knee radiographs when evaluating a patient for knee pain. This will be considered when assessing if the patient is eligible to participate given their pathology. This can be a new diagnosis or an already established diagnosis. The previous treatments that they have received will be noted in the patient charts while screened for eligibility.

Patients taking opioids only recently (less than 3 months) will be required to halt treatment at the time of study enrollment. Opioids don't have anti inflammatory properties so a washout period is not necessary. General patient demographics will be collected using the electronic medical record including: Age, Sex, BMI, Radiographic Osteoarthritis scale (Kellgren Lawrence), which will be put into database by the study investigators and co investigators.

Consent will be obtained by study personnel in the clinical office setting after meeting all study criteria and diagnosis of knee osteoarthritis based on exam and knee xrays. All patients diagnosed with knee osteoarthritis, and who are enrolled in the study, will be prescribed physical therapy that focuses on non-operative treatment such as low impact exercises and activity modification. The patients will not medicate with anti-inflammatory while enrolled in the study. Administration will follow a model of topical patch application which will consist of either the formulated CBD patch (35mg) or identical placebo patch. This patch will be applied to the arthritic knee directly central on the knee. In the event of patients with a diagnosis of bilateral knee OA, the patch will be placed on the knee that has visual analogue scale (VAS) >3 but <9. This patch will be placed daily for 24 hours and replaced each day. Including the initial enrollment visit, the patient will meet with the diagnosing orthopedic surgeon at various time points, and will also have remote check ins by study personnel to assess for adverse events and any issues they are having at 2, 4, and 8 weeks. The patient will have the patch for the first 4 weeks of the study followed by 4 weeks without patch which will conclude their participation at 8 weeks. The patients will all begin physical therapy as part of their routine clinical care within 1 week of beginning the study. During this time the patient will be distributed various surveys to measure patient outcomes. The investigators will be looking at pain as a primary endpoint using visual analogue scale with a 2 point difference deemed the minimal clinically important difference.

Subjects who are randomized to either group who have uncontrolled pain will be instructed to take a rescue medication, acetaminophen over the counter use Q 6 hours as needed will be allowed and recorded in a daily drug use diary which will be provided to them.

The patients will have contact information of the surgeon and residents to contact if any side effects are encountered. Compliance with patch use/application, side effects and adherence to physical therapy will also be recorded. Software with be used for both data collection and survey administration for confidential participation, which is a user-friendly HIPAA compliant service utilized by our health system. If the patient is unable to respond to the surveys via their phone app then hard copies of the survey will be given to them and collected by the investigator.

ELIGIBILITY:
Inclusion Criteria:

1. Age>18 years old
2. Osteoarthritis diagnosed radiographically as Kellgren Lawrence classification 2-4
3. Visual analogue scale greater than 3 but less than 9
4. Subject is able to provide written informed consent prior to any study procedures or interventions.
5. Ability, in the opinion of the investigator, to understand the nature of the study and comply with protocol requirements including compliance with scheduled visits, treatment plan, and any other study procedures outlined in this protocol.
6. Able to wear a patch for 24 hours a day
7. Able to participate in physical therapy

Exclusion Criteria:

1. Subject presents with a visual analogue scale score less than 4 or greater than 8.
2. Subject is Pregnant.
3. Patient has known recent substance abuse or dependence on alcohol (regularly consumes 3 or more alcoholic drinks per day), narcotic analgesics, tranquilizers, or opioids; in the judgement of the investigator within the past 3 years.
4. Subject has had prior surgery to the studied lower extremity within 6 months.
5. Subject has a known history of allergy to CBD or its derivatives
6. Subject has a known history of allergic, idiosyncratic, or serious adverse reactions to acetaminophen.
7. Patient had recent steroid injection to the studied knee within the last 3 months
8. Subject has an inability to be available for follow up
9. Any patients with prior liver pathology including, cirrhosis, hepatitis, Hepatic Carcinoma, or elevated liver function tests will be excluded from the study group. Patients with elevated baseline transaminase levels above 3 times the upper limit of normal, accompanied by elevations in bilirubin above 2 times the upper limits of normal.
10. Subjects with a medical disorder, condition or history such that could impair the subject's ability to participate or complete this study in the opinion of the investigator.
11. Patient has chronic opioid dependency (taking opioid's >3months), currently taking selective serotonin reuptake inhibitor or benzodiazepines.
12. Patient currently using CBD product and not willing to discontinue use 1 week prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-12 (Estimated); Study Completion 2024-02 (Estimated)

PRIMARY OUTCOMES:
Influence of CBD patch on pain for patients with knee osteoarthritis using Visual Analogue Scale. | 8 weeks.
  Efficacy of 35mg CBD Patch vs Placebo Patch on treatment of pain for patients with knee osteoarthritis assessed by a visual analogue scale using 0 as no pain and 10 as the worst pain. This will be collect at weeks 1, 2, 3, 4, and 8, where pain control method (CBD vs Placebo) is the between subjects' effect and week of treatment is the within subjects effect will be used to examine the association between pain control method and that outcome.

SECONDARY OUTCOMES:
Influence of CBD patch on physical and mental health for patients with knee osteoarthritis using the Short Form-12. | 8 weeks.
  The Short Form-12 (SF-12) will be used to asses physical functioning, physical health problems, limitations, emotional problems and global mental health. Two summary scores, a mental component score (MCS-12) and a physical component score (PCS-12), are reported as difference compared to the population average, measured in standard deviations. Each increment of 10 points above or below 50, corresponds to one standard deviation away from the average. Increasing scores correspond to positive physical (maximum 56.6)/mental health (maximum 60.8), decreasing scores correspond to negative physical (minimum 24.0)/mental (minimum 19.1) health.
Influence of CBD patch on quality of sleep for patients with knee osteoarthritis using the Pittsburgh Sleep Quality Index. | 8 weeks.
  The Pittsburgh Sleep Quality Index (measures quality and patterns of sleep) will be given prior to enrollment, and at weeks 1,2,3,4,8. Measures seven domains: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction over the last month. Scoring of the answers is based on a 0 to 3 scale, whereby 3 reflects the negative extreme.
Influence of CBD patch on physical function and emotional health for patients with knee osteoarthritis using the Brief Pain Inventory. | 8 weeks.
  Physical function will be measured by the activity sub dimension of the reactive dimension of the Brief Pain Inventory (BPI) (total of the scores for walking, general activity, and work items) Emotional function will be measured by the affective sub dimension of the reactive dimension of the BPI (Total of the scores for relations with others, enjoyment of life, mood, and sleep), on a 0 to 10 scale, where 10 is the negative extreme.
Influence of CBD patch on knee function and pain for patients with knee osteoarthritis using the Knee Injury and Osteoarthritis Outcome Score. | 8 weeks.
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) test will assess pain and function of the knee. Scores range from 0 to 100 with a score of 0 indicating the worst possible knee symptoms and 100 indicating no knee symptoms.
Safety Profile and Adverse Effects of CBD patch | 8 weeks.
  The safety of the CBD patch will be assessed by a 15 item questionnaire of the most commonly reported adverse events of cannabinoids in prior literature. Additional adverse reactions reported by patients or observed by the investigator will be noted and scored.
  Scoring of the severity is based on a 0 to 3 interval scale (corresponding to none, mild, moderate, severe), whereby 3 reflects the negative extreme. The patients will be proactively assessed at 2, 4, and 8 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Vijay Rasquinha, MD, Principal Investigator — Northwell Health; Robert Duarte, MD, Study Director — Northwell Health
Locations (1):
- Northwell Health Orthopedic Institute at Great Neck, New Hyde Park, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baer PA, Thomas LM, Shainhouse Z. Treatment of osteoarthritis of the knee with a topical diclofenac solution: a randomised controlled, 6-week trial [ISRCTN53366886]. BMC Musculoskelet Disord. 2005 Aug 8;6:44. doi: 10.1186/1471-2474-6-44. PMID 16086839
- [Background] Martin-Santos R, Crippa JA, Batalla A, Bhattacharyya S, Atakan Z, Borgwardt S, Allen P, Seal M, Langohr K, Farre M, Zuardi AW, McGuire PK. Acute effects of a single, oral dose of d9-tetrahydrocannabinol (THC) and cannabidiol (CBD) administration in healthy volunteers. Curr Pharm Des. 2012;18(32):4966-79. doi: 10.2174/138161212802884780. PMID 22716148
- [Background] Haney M, Malcolm RJ, Babalonis S, Nuzzo PA, Cooper ZD, Bedi G, Gray KM, McRae-Clark A, Lofwall MR, Sparenborg S, Walsh SL. Oral Cannabidiol does not Alter the Subjective, Reinforcing or Cardiovascular Effects of Smoked Cannabis. Neuropsychopharmacology. 2016 Jul;41(8):1974-82. doi: 10.1038/npp.2015.367. Epub 2015 Dec 28. PMID 26708108
- [Background] Babalonis S, Haney M, Malcolm RJ, Lofwall MR, Votaw VR, Sparenborg S, Walsh SL. Oral cannabidiol does not produce a signal for abuse liability in frequent marijuana smokers. Drug Alcohol Depend. 2017 Mar 1;172:9-13. doi: 10.1016/j.drugalcdep.2016.11.030. Epub 2016 Dec 14. PMID 28088032
- [Background] Philpott HT, O'Brien M, McDougall JJ. Attenuation of early phase inflammation by cannabidiol prevents pain and nerve damage in rat osteoarthritis. Pain. 2017 Dec;158(12):2442-2451. doi: 10.1097/j.pain.0000000000001052. PMID 28885454
- [Background] Malfait AM, Gallily R, Sumariwalla PF, Malik AS, Andreakos E, Mechoulam R, Feldmann M. The nonpsychoactive cannabis constituent cannabidiol is an oral anti-arthritic therapeutic in murine collagen-induced arthritis. Proc Natl Acad Sci U S A. 2000 Aug 15;97(17):9561-6. doi: 10.1073/pnas.160105897. PMID 10920191
- [Background] Hammell DC, Zhang LP, Ma F, Abshire SM, McIlwrath SL, Stinchcomb AL, Westlund KN. Transdermal cannabidiol reduces inflammation and pain-related behaviours in a rat model of arthritis. Eur J Pain. 2016 Jul;20(6):936-48. doi: 10.1002/ejp.818. Epub 2015 Oct 30. PMID 26517407
- [Background] Xiong W, Cui T, Cheng K, Yang F, Chen SR, Willenbring D, Guan Y, Pan HL, Ren K, Xu Y, Zhang L. Cannabinoids suppress inflammatory and neuropathic pain by targeting alpha3 glycine receptors. J Exp Med. 2012 Jun 4;209(6):1121-34. doi: 10.1084/jem.20120242. Epub 2012 May 14. PMID 22585736
- [Background] Lodzki M, Godin B, Rakou L, Mechoulam R, Gallily R, Touitou E. Cannabidiol-transdermal delivery and anti-inflammatory effect in a murine model. J Control Release. 2003 Dec 12;93(3):377-87. doi: 10.1016/j.jconrel.2003.09.001. PMID 14644587
- See also: Topical treatments for osteoarthritis of the knee - Database of Abstracts of Reviews of Effects (DARE): Quality-assessed Reviews - NCBI Bookshelf — https://www.ncbi.nlm.nih.gov/books/NBK73645/